CLINICAL TRIAL: NCT06526546
Title: ADVENT Trial Long Term Outcomes Evaluating Atrial Fibrillation Progression (ADVENT LTO Study)
Brief Title: ADVENT Trial Long Term Outcomes Evaluating Atrial Fibrillation Progression Study
Acronym: ADVENT LTO
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PF116
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; Pulsed Field Ablation; Cardiovascular Heart Diseases; Antiarrhythmic Anticoagulation; Cardiac monitor; Atrial Fibrillation; Atrial Flutter; Atrial Tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The (ADVENT LTO) is an observational, non-significant risk study to assess the progression of atrial fibrillation in subjects who received ablation treatment with either the FARAPULSE Pulsed Field Ablation System or thermal ablation in the ADVENT Trial.

DETAILED DESCRIPTION:
This study is an observational, non-significant risk study. Subjects who participated in the FARAPULSE ADVENT Trial (NCT04612244) will be approached for participation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria may be given consideration for inclusion in this clinical investigation.
* Subjects who were enrolled, randomized and treated for paroxysmal atrial fibrillation, classified as Modified Intention-to-Treat subjects, and completed the 12-Month Follow-Up in the FARAPULSE ADVENT Trial (CIP CS0934; NCT04612244).
* Subjects or legally authorized representatives who are willing and capable of providing informed consent.
* Subjects who are willing to comply with the protocol requirements.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study eligibility criteria are defined below. Subjects who became deceased after completion of the ADVENT Trial will remain eligible for chart review data upon consent of a legally authorized representative (LAR). Subjects unable to complete the 7-day Holter monitor may consent to participate in the chart review portion only.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Chronic success in ADVENT Trial treated subjects compared between treatment groups. | 90 day-3 years
  Occurrence of any of the following between the end of the Blanking Period (Day 90) in the ADVENT Trial through completion of follow-up in the ADVENT LTO study:
  Detectable AF, AFL+, or AT
  * ≥ 30 seconds in duration as adjudicated within the ADVENT Trial
  * Investigator assessed ≥ 30 seconds in duration from any approved clinical recording devices considered standard of care* at the study center post-ADVENT Trial completion
  * ≥ 30 seconds in duration recorded on the Holter monitor collected during the ADVENT Trial and the 3-4 Year Holter Monitor.
  * ≥ 10-second of continuous AF, AFL or AT documented on any 12-lead ECG
  Any Cardioversion for AF, AFL, or AT
  Re-ablation for AF, AFL, or AT

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (25):
- United States (25):
  - Grandview Medical Center, Birmingham, Alabama
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Mills Peninsula Health Services, Burlingame, California
  - Scripps Memorial Hospital, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital, Atlanta, Georgia
  - St. Lukes Idaho Cardiology Associates, Boise, Idaho
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Mount Sinai, Icahn School of Medicine, New York, New York
  - Northwell Health, New York, New York
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Presbyterian University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Pinnacle Health at Harrisburg Hospital, Wormleysburg, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Thomas Research Institute, LLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Virginia Commonwealth University Health System, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
No requests for study data have been made at this time, however Boston's Scientific's policy on data sharing can be found at http://www.bostonscientific.com/en-US/data-sharing-requests.html

REFERENCES:
- [Derived] Reddy VY, Gerstenfeld EP, Mountantonakis SE, Patel C, Ellenbogen KA, Harding JD, Gibson DN, Natale A, Waks JW, Calkins H, Gupta SK, Woods CE, Whang W, Daccarett M, Cuoco FA, Delurgio DB, Richards E, Martens MD, Sutton B, Mansour M; ADVENT-LTO Study Investigators. Pulsed Field versus Conventional Thermal Ablation for Paroxysmal Atrial Fibrillation: 4-Year Outcomes in the ADVENT-LTO Study. Nat Med. 2026 Feb 6. doi: 10.1038/s41591-026-04246-4. Online ahead of print. PMID 41652117